CLINICAL TRIAL: NCT05412732
Title: Study for the Clinical Validation of a New Biomarker to Determine Predisposition to Infections in Patients With Acute Myocardial Infarction.
Brief Title: Study for the Validation of a New Biomarker to Determine Predisposition to Infections in Patients With Acute Myocardial Infarction.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Collaborators: Crazy Science & Business S.L. (Unknown)
Responsible Party: Sponsor
Other Study IDs: BIOMIN-001
Record Dates: First submitted 2022-05-19; First posted 2022-06-09 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Infections in Acute Myocardial Infarction Patients

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — This clinical study aims to demonstrate, based on PCR analysis of a patient's blood sample, that levels of a mitochondrial DNA-based biomarker (mitoDNA) is able to predict the risk of infection for patients who have suffered Acute Myocardial Infarction (AMI).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group A low risk of infection
  Interventions: Other: prospective biomedical research study
- group B high risk of infection
  Interventions: Other: prospective biomedical research study

INTERVENTIONS:
Other: prospective biomedical research study — A prospective biomedical study, in which a comparison will be made of the outcome of a specific disease (in this case, AMI).

SUMMARY:
Prospective biomedical research study

DETAILED DESCRIPTION:
The aim is to validate a new biomarker, based on the levels of DNAmit present in blood, to assess the predisposition of an individual to suffer an infection. To validate this hypothesis, the DNAmit levels of patients with myocardial infarction will be analysed and their relationship with the probability of these patients developing an infectious process or not.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have suffered AMI or cardiorespiratory arrest after AMI, have been admitted to hospital within the first 24 hours of the event and are required to be admitted to any Critical Care Unit. In addition, one of the following criteria must be met:

  1. Symptoms of cardiac ischaemia.
  2. New ischaemic patterns in the ECG.
  3. Development of pathological QW waves on the ECG.
  4. Obvious suspicion or loss of myocardial viability or new abnormal motility regions in a pattern consistent with ischaemic pathology.
  5. Intracoronary thrombus detected on angiography or autopsy. 2. They must be of legal age, have read the Patient Information Sheet (HIP) and have signed the Informed Consent (IC).

     Depending on the group in which they are to be classified, patients must meet specific inclusion criteria:

     Group A: Patients who have suffered MI (myocardial infarction), are in the CRITICAL UNIT and their DNAmit values are below 0.25-105 copies.

     Group B: Patients who have suffered an MI, are in the CRITICAL UNIT and their mtDNA values are above 0.25-105 copies.

     Exclusion Criteria:

     Patients who meet any of the following criteria shall not be eligible for inclusion in the clinical trial:
     1. Chronic inflammatory diseases
     2. Transplantation of any organ (except cornea).
     3. Patients receiving or who have received in the last 3 months anti-inflammatory, immunosuppressive or biological treatment targeting the immune system (TNF blockers, anakinra, rituximab, abatacept or tocilizumab), except NSAIDs and colchicine.
     4. Patients with overt and/or severe immunocompromise
     5. History of chronic kidney or liver disease (dialysis or creatinine clearance < 30%).
     6. Decompensated diabetes
     7. Active tumour process. Patients considered to be in complete remission may be included in the study.
     8. Major surgical intervention (in the 3 MONTHS PRIOR to inclusion in the study).
     9. Pregnancy, childbirth or breastfeeding in the last 3 months.
     10. Symptomatic patients with type IV heart failure (NYHA).
     11. Life expectancy of less than 3 months.
     12. Long-term urinary catheter or vascular catheter wearers

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is aimed at those patients who have suffered an AMI or OUT-OF-HOSPITAL CARDIORRESPIRATORY ARREST and are admitted to the Critical Care Unit.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-07-21 (Actual); Primary Completion 2022-07-21 (Estimated); Study Completion 2023-07-21 (Estimated)

PRIMARY OUTCOMES:
Clinical validation of the presence of elevated mitochondrial DNA levels as a prognostic biomarker of infection risk in AMI patients | 18-30 hours
  Level of circulating DNAmit

SECONDARY OUTCOMES:
Correlating mitochondrial DNA levels with the patient's "immune" tolerant status | 18-30 hours
  Refractory state of circulating monocytes/macrophages [pg/mL]
To determine the relationship between ADNmit levels and infarct location | 0-24 hours
  Infarct location (anterior or non-anterior)
To determine the relationship between ADNmit levels and Left Ventricular Ejection Fraction | 0-24 hours
  LVEF [%]
To determine the relationship between ADNmit levels and ultrasensitive troponin I | 0-24 hours
  ultrasensitive troponin I [pg/mL]
To determine the relationship between ADNmit levels and GRACE Score | 0-24 hours
  GRACE Score [numerical values that determine risk of death: 0-258]

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario La Paz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No